CLINICAL TRIAL: NCT06502847
Title: The Role of Breastmilk and Serum Exosome Profile in Prediction of the Severity and Treatment Requirement of Neonatal Jaundice Due to ABO Incompatibility
Brief Title: The Role of Breastmilk and Serum Exosomes in Neonatal Jaundice Due to ABO Incompatibility
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Seda Yilmaz Semerci, Assoc Prof, Health Institutes of Turkey
Other Study IDs: 43057
Record Dates: First submitted 2024-07-09; First posted 2024-07-16 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Neonatal Jaundice From Other Specified Causes; ABO Incompatibility; ABO Hemolytic Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Case ABO1: Newborns who receive treatment due to the ABO Incompability will be included in this group.
  Interventions: Other: Exosome profile study
- Case ABO2: Newborns who have the ABO Incompability, but do not require treatment will be included in this group.
  Interventions: Other: Exosome profile study
- Control: Healthy newborns without any disease or health condition will be included in this group
  Interventions: Other: Exosome profile study

INTERVENTIONS:
Other: Exosome profile study — Neonatal serum and maternal exosome profiles will be studied in all groups.

SUMMARY:
Neonatal jaundice is a major global health issue that can lead to serious complications and even death if not promptly treated. ABO incompatibility is a common cause of pathological neonatal jaundice, but there are currently no specific tests to predict its severity or progression. This project aims to study the role of exosomes in the diagnosis and treatment of newborn jaundice, focusing on their impact on infants with ABO incompatibility. The study will take place at a reference neonatal intensive care unit, involving 45 infants. Serum and breast milk samples will be collected and analyzed to determine any relationships and possible correlations.

ELIGIBILITY:
Inclusion Criteria:

* Newborns who are needed treatment for neonatal jaundice due to ABO incompatibility
* Newborns who are admitted to the study center due to ABO hemolytic disease
* Newborns with ABO incompatibility
* Healthy newborns
* Healthy mothers

Exclusion Criteria:

* Lack of informed consent
* Congenital abnormalities
* Maternal Liver diseases
* Neonatal liver diseases
* Sepsis
* Neonatal jaundice due to the causes other than ABO incompatibility
* Acute or chronic disease state in newborn
* Maternal acute or chronic disease
* Medication or substance use effecting liver functions

Max Age: 28 Days | Sex: All
Age Groups: Child
Study Population: It is planned to include a total of 45 babies in the study, including healthy babies (n=15) in the first group, babies who developed jaundice due to ABO incompatibility but did not need treatment (n=15) in the second group, and babies who developed jaundice due to ABO incompatibility and needed treatment (n=15) in the third group.
Sampling Method: Non-Probability Sample
Enrollment: 338 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Number of the participant who Need for Treatment | 12 months
  Association between the serum and breastmilk exosome and need for treatment due to ABO incompability

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences Istanbul KSS Training and Research Hospital, Istanbul, Kucukcekmece, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No